CLINICAL TRIAL: NCT04464850
Title: Effects Intravenous Iron and Oral Iron Therapy on Erythropoietin Dose in Maintenance Hemodialysis Patients: An Open-label, Randomized, Controlled Study
Brief Title: Intravenous Versus Oral Iron Therapy in Hemodialysis Patients
Acronym: IVO-IRON
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kajohnsak Noppakun, Assistant Professor of Medicine, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MED-2563-07092
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Hemodialysis Complication; Anemia; Iron Deficiency Anemia
Keywords: Iron therapy; Hemodialysis; Iron status; Epoetin dose; Intravenous iron; Oral iron
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency | interventions — Ferric Oxide, Saccharated; Iron; ferrous fumarate; Folic Acid

STUDY DESIGN:
Intervention Model Description: Maintenance hemodialysis patients who are eligible to enrol into the study according to inclusion and exclusion criteria will be start with 2-week run-in period before randomization. During this run-in period, all iron supplements that patients receive including oral and intravenous iron will be discontinued.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous iron (Experimental): Iron sucrose 200 mg every 2 weeks Folic acid 5 mg/day B6 10 mg/day
  Interventions: Drug: Intravenous iron
- Oral iron (Active Comparator): Ferrous fumarate 600 mg/day Folic acid 6.5 mg/day B6 15 mg/day
  Interventions: Drug: Oral iron

INTERVENTIONS:
Drug: Intravenous iron — Iron sucrose will be given by continuous infusion for 1 hour during the last 1 hour of dialysis session. Iron sucrose will be given for 24 weeks during study period.
  Serum ferritin will be monitored at 4, 12, and 24 weeks after randomization.
  The dosage of intravenous iron will be adjusted according to serum ferritin levels as follows.
  Serum ferritin <500 mg/dl: iron sucrose 100 mg every 2 weeks Serum ferritin 500-800 mg/dl: iron sucrose 100 mg every 4 weeks Serum ferritin >800 mg/dl: discontinue iron sucrose
  Other Names: Venofer, Encifer
  Arms: Intravenous iron
Drug: Oral iron — 1 tablet, three times a day, of iron fumarate will be prescribed for 24 weeks of study period.
  The dosage of iron fumarate will be adjusted according to serum ferritin levels as follows.
  Serum ferritin will be monitored at 4, 12, and 24 weeks after randomization.
  Serum ferritin <500 mg/dl: iron fumarate 200 mg three times daily Serum ferritin 500-800 mg/dl: iron fumarate 200 mg once daily Serum ferritin >800 mg/dl: discontinue iron fumarate
  Other Names: Ferli-6 (ferrous fumarate 200 mg, folic acid 0.5 mg, B6 5 mg)
  Arms: Oral iron

SUMMARY:
This study is aim to compare the efficacy of intravenous versus oral iron therapy regarding the hemoglobin levels, iron status and erythropoietin dosage in maintenance hemodialysis patients

DETAILED DESCRIPTION:
Run-in phase: All eligible patients will enter run-in phase for 2 weeks. In this phase, all oral therapy that patients received before enrolment into the study will be discontinued.

Masking: Opened label

Allocation: Block of four randomization into 2 treatment arms: intravenous iron and oral iron

Safety criteria: Study participants who meet the following criteria will be discontinued from the study. All patients data will be analyzed according to intention-to-treat principles.

* Hemoglobin levels < 6.0 g/dl
* Packed red cells transfusion is required
* Serum ferritin >1,000 md/dl

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Hemodialysis for at least 3 months
* Hemoglobin levels between 8 and 11.5 g/dl inclusive
* Transferrin saturation (TSAT) <50% and ferritin <800 mg/dl
* Stable dose of epoetin of any types and iron therapy for at least 1 month

Exclusion Criteria:

* History of iron allergy
* Pregnant or lactating women
* Patients with known hematologic disorders other than anemia of renal disease and iron deficiency anemia
* Patients with hemoglobinopathy e.g., thalassemia
* Patients with iron overload or hemochromatosis
* Patients with gastrointestinal hemorrhage during 6 months before enrolment in to the study
* Patients with current severe infection
* Patients with any malignancies
* Patients with severe psychiatric illness
* Patients with any other medical condition which, in the Investigator's judgment, may be associated with increased risk to the subject or may interfere with study assessments or outcomes
* Patients who currently receive medications that can altered gastrointestinal absorption of oral iron e.g., aluminum carbonate, aluminum hydroxide, chloramphenicol, dimercaprol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes of epoetin dose | 24 weeks after randomization
  Hemoglobin levels will be monitored and epoetin dose will be adjusted according to hemoglobin levels at 4, 12, 24 weeks after randomization.
  Protocols for epoetin dose adjustments are shown as follow. Hemoglobin levels (g/dl) Epoetin dose adjustment <9.0 Increased by 50% 9.0 to <10.0 Increased by 25% 10.0 to <11.5 No change 11.5 to <12.5 Decreased by 25%
  * 12.5 Decreased by 50%

SECONDARY OUTCOMES:
Hemoglobin levels | 4, 12, 24 weeks after randomization
  Levels of hemoglobin concentration
Erythropoietin resistance index | 4, 12, 24 weeks after randomization
  Erythropoietin resistance index is calculated as the mean weekly epoetin dose per kg body weight divided by the average hemoglobin level
Major cardiovascular events (MACE) | 24-week period after randomization
  Major adverse cardiovascular events (MACE) is defined as a composite of nonfatal stroke, Nonfatal myocardial infarction, and cardiovascular death
Unscheduled hospitalization | 24-week period after randomization
  Numbers of any hospitalizations that is not planned
Hospitalization due to infections | 24-week period after randomization
  Numbers of any hospitalizations that is caused by infections
C-reactive protein (CRP) | 4, 12, 24 weeks after randomization
  Serum levels of high sensitivity c-reactive protein
The kidney disease quality of life (KDQOL) instrument | 4, 12, 24 weeks after randomization
  Quality of life will be assessed by the kidney disease quality of life (KDQOL) instrument
Quality of life will be assessed by EQ-5D-5L (EuroQol - 5 Dimensions - 5 Levels) | 4, 12, 24 weeks after randomization
  EQ-5D-5L is the instrument used to evaluate health-related quality of life states in adults, consisting of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression), each of which has five severity levels
Cost-effectiveness of iron therapy | 4, 12, 24 weeks after randomization
  The cost of iron therapy compared with the cost of epoetin

CONTACTS AND LOCATIONS:
Overall Officials: Kajohnsak Noppakun, MD, Principal Investigator — Instructor, Division of Nephrology, Department of Internal Medicine
Locations (1):
- Chiang Mai University Hospital, Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No
Request for individual participant data (IPD) has to be submitted to the Institutional Review Board (IRB) of Faculty of Medicine, Chiang Mai University, Chiang Mai, THAILAND.